CLINICAL TRIAL: NCT05092204
Title: Prevalence and Risk Factors of Dermatoporosis in Patients Over 75 Years of Age Hospitalized in Reeducation
Acronym: Dermatoporose
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210431
Record Dates: First submitted 2021-05-14; First posted 2021-10-25 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2021-10

CONDITIONS: Dermatoporosis
Keywords: Skin aging; Dermatoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patient in SSR geriatric service

SUMMARY:
The term dermatoporosis, by analogy to osteoporosis, was proposed by Professor Saurat to define all the manifestations linked to skin aging leading to fragility and skin failure. With age, the gradual disappearance of hyaluronic acid and its CD44 cell receptor leads to the degeneration of the extracellular matrix and then to the loss of the protective mechanical functions of the skin. It thus appears an alteration of the viscoelasticity of the skin. The most common skin manifestations of dermatoporosis are mainly located on the upper limbs. Several clinical manifestations characterize dermatoporosis: skin atrophy, senile purpura, stellate pseudo-scars, delayed healing and finally dissecting skin hematoma. There are 4 evolutionary stages of dermatoporosis described by Professor Saurat and by Doctor Kaya, in 2007: Stage 1: strong thinning of the skin with senile purpura and stellate pseudo-scars. Stage 2: manifestations of the previous stage and small, localized skin lacerations resulting from a cleavage between the dermis and the epidermis. Stage 3: more and larger skin lacerations with a noticeable delay in healing Stage 4: the progression of the lesions described above leads to the formation of dissecting skin hematomas which may progress to skin necrosis. (Saurat JH Dermatoporosis - the functional side of skin aging. Dermatology 2007 and Kaya G, dermatoporosis: A chronic cutaneous insufficiency / fragility syndrome. Clinicopathological features, mechanisms, prevention and potential treatments. Dermatology 2007).

A study by Mengeaud et al found a significant association between severe renal failure and dermatoporosis. Two studies, one in Toulouse and the other in Finland, looked at the prevalence and risk factors of dermatoporosis in patients over 60 years of age. The observational study on 202 patients over 60 years old in Toulouse shows a prevalence of 32%, with preferentially localization on the upper limbs. Stage 1 is the most common. Multivariate statistical analyzes show that dermatoporosis is significantly associated with the use of local and oral corticosteroids, anticoagulants, and chronic renal failure. On the other hand, it has not been shown to be associated with diabetes and the patient's sun exposure.Another study, dating from 2018 also found that kidney failure, taking antiaggregants and anticoagulants, corticosteroid therapy (local or systemic) are risk factors for dermatoporosis. However, no study has been carried out on a geriatric population, and the association between phototype, sun exposure and dermatoporosis has to our knowledge never been systematically investigated in the few studies conducted.

DETAILED DESCRIPTION:
This study will allow us to know the prevalence and the risk factors of dermatoporosis in a poorly understood geriatric population. No study on the subject in patients over 75 years in the literature. We will be interested in collecting on the observations of patients recorded in Orbis (Initial medical assessment and evolution), in particular if the patient has chronic renal failure, is diabetic, has anticoagulants, antiaggregants or corticosteroids as a background treatment.

Main objective To assess the prevalence of dermatoporosis in patients over 75 years of age hospitalized in reeducation. Secondary objectives: Investigate risk factors for dermatoporosis - Evaluate the prevalence of complications of dermatoporosis

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient in SSR
* Over 75 years old patient

Exclusion Criteria:

* Refusal of participation

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patient in SSR over 75 years old.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Presence or absence of dermatoporosis | From admission to discharge, up to 1 month
  Presence or absence of dermatoporosis in geriatric patients hospitalized in the CRH

SECONDARY OUTCOMES:
Measurement of phototype | At admission, Day 1
  Measurement of phototype as a risk factors for dermatoporosis
Childhood sun exposure Measurement of phototype | At admission, Day 1
  Childhood sun exposure as a risk factors for dermatoporosis
Lifetime sun exposure Measurement of phototype | At admission, Day 1
  Lifetime sun exposure as a risk factors for dermatoporosis
Complications of dermatoporosis: | At admission, Day 1
  Complications of dermatoporosis: dissecting hematoma, skin tear on clinical examination and in history

CONTACTS AND LOCATIONS:
Overall Officials: Hester COLBOC, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital ROTSCHILD, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided